CLINICAL TRIAL: NCT05834296
Title: Randomized, Double-blind, Placebo-controlled, Parallel-group, Phase 1/2a Study to Assess Safety, Tolerability & Efficacy of Autologous Beta-Amyloid Mutant Peptide-pulsed Dendritic Cells in Subjects With Mild-to-Moderate Alzheimer's Dementia
Brief Title: Study in Subjects With Mild-to-Moderate Alzheimer's Dementia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alzamend Neuro, Inc. (Industry)
Collaborators: bioRASI, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALZN002-01
Record Dates: First submitted 2023-02-22; First posted 2023-04-28 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Each cohort will have 10 total subjects randomized in a 7:3 ratio (active:placebo). Subjects will be randomly allocated to treatment groups based on a central computer-generated randomization scheme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): ALZN002 (autologous DCs pulsed with E22W mutant peptide).
  Interventions: Biological: ALZN002 (autologous DCs pulsed with E22W mutant peptide).
- Placebo (Placebo Comparator): Saline ID and IV administrations.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: ALZN002 (autologous DCs pulsed with E22W mutant peptide). — The cellular immunotherapy product consists of autologous dendritic cells (DCs) pulsed with a novel amyloid-beta peptide (Aβ1 42) containing a mutation at position 22 from glutamic acid to tryptophan (E22W). This mutation produces novel CD4+ T cell epitopes specific for the mutant E22W peptide that can facilitate an anti-Aβ1-42 antibody response. The activated E22W peptide specific CD4+ T cells license Aβ1-42-specific B cells to secrete anti Aβ1-42 antibodies, resulting in systemic reduction of amyloid and reduction or slowed accumulation of amyloid plaques in the brain.
  Arms: Active
Drug: Placebo — Saline
  Arms: Placebo

SUMMARY:
ALZN002-01 is a first-in-human, randomized, double-blind, placebo-controlled, parallel-group, phase 1/2a study of autologous amyloid beta mutant peptide-pulsed dendritic cells (ALZN002) in subjects with mild-to-moderate dementia of the Alzheimer's type.

DETAILED DESCRIPTION:
ALZN002-01 is a first-in-human, randomized, double-blind, placebo-controlled, parallel-group, phase 1/2a study. The primary purpose of this study is to assess the safety and tolerability of multiple ascending doses of ALZN002 compared with that of placebo in subjects with mild to moderate dementia of the Alzheimer's type (AD) and to determine the optimal dosage of ALZN002 that allows for induction of anti-amyloid-beta (Aβ) antibody responses while maintaining safety. The overall goal of this study is to determine an appropriate dose to use in a larger phase 2b study (ALZN002-02) where efficacy is the primary study purpose.

ELIGIBILITY:
Inclusion Criteria:

Potential study subjects must satisfy the following criteria to be randomized in the study:

1. Age ≥60 and ≤85 years with no restrictions on gender, race, or ethnicity.
2. Able and willing to give informed consent and adhere to study requirements, including testing for cognitive and functional abilities.
3. Confirmation of AD at Screening based either on a positive amyloid PET obtained at Screening or based on historical positive amyloid PET taken within 6 months prior to the screening visit consistent with AD. If historical amyloid PET imaging is used for inclusion

   1. there should be no clinically significant change in the subject's symptoms and cognitive abilities within the 6 months prior to Screening.
   2. The quality and accuracy of the historical positive amyloid PET needs to be confirmed by the central imaging center
4. Willing and able to have amyloid PET taken at Screening (if no historical adequate amyloid PET within 6 months of Screening is available) to confirm AD and at Week 31 and Week 143 as a potential efficacy measure.
5. Willing and able to have magnetic resonance imaging (MRI) taken at Screening, at 1 year (Week 55) and 2 years (Week 101) after the 3rd dose, and at 1 year after the 10th dose (Week 143/EOS) as potential safety measures.
6. Males (non-vasectomized and vasectomized) must agree to use barrier contraception during the study until 30 days after the last dose of the study investigational treatment.
7. Females must meet one the of the following criteria:

   a. Either is of childbearing potential and agrees to use an acceptable contraceptive method. Acceptable contraceptive methods include:

   i. Abstinence from heterosexual intercourse from the Screening visit through to at least 30 days after the last dose of the study investigational treatment

   ii. One of the following highly-effective contraceptive methods, used from at least 28 days prior to the Screening visit through to at least 30 days after the last dose of the study investigational treatment:
   * Systemic contraceptive (combined birth control pills, injectable/implant/insertable hormonal birth control products, or transdermal patch)
   * Intrauterine device (with or without hormones)
   * Male condom used with male partner vasectomized at least 6 months prior to the Screening visit

   iii. One of the following double-barrier contraceptive methods, used from the Screening visit through to at least 30 days after the last dose of the study investigational treatment:
   * Male condom used simultaneously with diaphragm plus spermicide
   * Male condom used simultaneously with cervical cap plus spermicide

   Or

   b. Is of non-childbearing potential, defined as surgically sterile (ie, has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation), or is in a postmenopausal state (ie, at least 1 year without menses, not attributable to another cause, prior to the Screening visit)
8. In the event that the subject requires a study partner, he/she must be reliable and will provide written informed consent to participate and be in frequent contact with the participant. The study partner must be familiar with the subject's overall function and behavior, such as day-to-day activities and cognitive abilities.
9. Able to speak, read, and write (for cognitive testing).
10. Clinical diagnosis of probable or possible AD based on National Institute on Aging - Alzheimer's Association (NIA-AA) criteria by a qualified clinician.
11. Clinical diagnosis of at least mild dementia according to the CDR Global Score of 0.5 to 2 at screening and Baseline
12. Mini-Mental State Examination (MMSE) score of 14 - 26 and ADAS-cog11 score greater than 12 at screening and Baseline.
13. Willing and able to undergo leukapheresis as needed.
14. Consent to undergo d HLA geno-typing and PaxGene RNA.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from participating in the study:

1. Prior immunotherapies and specifically therapies that may elicit T cell or antibody responses to Aβ, whether investigational or approved by the FDA, for AD or other conditions.
2. Central nervous system-related exclusions:

   1. Delirium, non-AD dementia or cognitive impairment, or other encephalopathies.
   2. Subjects with major psychiatric disorder such as schizophrenia, bipolar disorder or major depressive disorder, or has current alcohol or substance abuse based on psychiatric consultation at Screening visit.
   3. Neuropsychiatric Inventory (NPI-Q) total score ≥14 or score ≥4 in any NPI domain (clinically significant neuropsychiatric symptoms). Apathy score ≥4 acceptable.
   4. At risk for suicide in the opinion of the investigator or the subject answers "yes" to "Suicidal Ideation" Item 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) (at the time of evaluation) at the screening visit or attempted suicide within the last 2 years.
   5. Modified Hachinski Scale10 score >4 or evidence of stroke within the past 5 years.
   6. Neuroimaging exclusions by history or entry criteria: Arteriovenous malformation, brain mass, suggestive changes of cerebral amyloid angiopathy (CAA), aneurysms, or other changes that increase risk of hemorrhage, multiple cerebral macrohemorrhages, or other cerebrovascular complications as deemed by the Principal Investigator and/or the Safety Adjudication Committee that might account for cognitive symptoms.
   7. MRI-related exclusion criteria: >4 lacunar infract, Grade III white matter hyperintensities (Fazekas scale), intracranial mass, evidence of normal pressure hydrocephalus or other anatomical findings that might affect safety or causes of cognitive impairments, and any contraindications for MRI scanning, including implanted metallic devices (eg, non MRI safe cardiac pacemaker or neurostimulator; some artificial joints; metal pins; surgical clips; or other implanted metal parts), or claustrophobia or discomfort in confined spaces.
   8. History of moderate or more severe traumatic brain injury in the 2 years prior to signing the consent to participate in the study.
   9. History of brain tumor, subdural hematoma, or other clinically significant (in the judgment of the investigator) space-occupying lesion on MRI.
   10. History of seizure disorder.
   11. Contraindications for PET scanning or any protocol testing procedure.
3. Systemic related exclusions:

   1. Known autoimmune disease (properly treated hypothyroidism and stable rheumatoid arthritis allowed), biomarkers exceeding 1:80 for antinuclear antibodies, 20 IU/mL (or 1:80) for rheumatic factor, 26 AU/mL for antineutrophil cytoplasmic antibodies; or history of allergic reaction to any related product of infused cells.
   2. Current malignancy, with the exception of non-invasive (stage 0 or stage 1) basal and squamous cell carcinoma with planned excision. Subjects with a prior successfully treated malignancy and a sufficient follow-up to exclude the likelihood of recurrence may be enrolled at the discretion of the Principal Investigator.
   3. History of or current HIV, HBV, or HCV (unless subjects who test positive for hepatitis C antibody are in remission with sustained virologic response, as evidenced by undetectable HCV RNA level using a sensitive assay ≥12 weeks after completion of HCV therapy).
   4. Elevated C-reactive protein (>5.0 mg/L) using a high sensitivity test.
   5. Fever, signs or symptoms of active illness or infection, or a diagnosed infectious disease.
   6. Immunizations within 4 weeks of the leukapheresis or investigational treatment (ALZN002 or placebo) administrations.
   7. Recent (past 8 weeks) donation of blood or loss of blood (>400 cc).
   8. Insulin-dependent diabetes mellitus
4. The following medications are excluded with the noted exceptions:

   1. Initiation of cholinesterase inhibitors, memantine HCl, or other drugs for the treatment of cognitive loss within 60 days of Screening, unless the dose is stable for >60 days prior to Screening and is expected to remain stable throughout the study participation
   2. Administration of diphenhydramine and/or acetaminophen are prohibited pre- and/or post-infusion except if, in the opinion of the Investigator on a case-by-case basis in response to individual subject infusion reaction adverse event(s), these drugs are judged to be appropriate for immediate treatment of adverse experiences and/or prophylactically prior to subsequent doses. Also, if adjudicated by the Sponsor's Expert Panel and Safety Adjudication Committee as appropriate, conditions of routine use of these drugs can be deployed during the study
   3. Treatment with coumarins/indandiones, factor Xa inhibitors, heparins, direct thrombin inhibitors, and aspirin, except low-dose (81 mg) aspirin for cardio-protection
   4. Benzodiazepines are permitted as a sleep aid only if taken at a stable dose for at least 60 days prior to Screening and the subject intends to continue to maintain the same regimen
5. Initiation of medications that could cause or worsen cognitive impairment (ie, anticholinergic medications, tricyclic antidepressants, antipsychotic medications, and anticonvulsant medications).
6. Initiation of systemic corticosteroid exposure or any other immunotherapies, regardless of indication, within 3 weeks prior to or after investigational treatment (ALZN002 or placebo) administrations, and immunizations within 4 weeks of the leukapheresis procedure or investigational treatment administrations.
7. Clinical laboratory exclusions:

   1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2 x upper limit of normal (ULN)
   2. Total bilirubin >1.5 x ULN unless Gilbert's syndrome
   3. Estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m2 (CKD-EPI 2022 formula)
   4. HbA1c >6.5%
   5. Hemoglobin <11.0 for males and <9.5 for females, use of red blood cell related medications/treatments (erythropoietin) within 2 years, history of or current bone marrow disease or myelodysplastic syndromes.
   6. Thyroid stimulating hormone >1.5 x ULN or <0.8 x lower limit of normal (LLN)
8. Electrocardiogram findings of ischemia or infarct, complete bundle branch blocks, symptomatic arrhythmias or predominantly non-sinus-conducted rhythm, QTcF >460 msec males or >480 msec females
9. Positive urine drug screen for controlled substances, including tetrahydrocannabinol or controlled substance(s) for which the subject does not have a valid prescription. Subjects taking non tetrahydrocannabinol (THC) containing cannabidiol products will not be excluded unless the urine drug screen is positive for THC.
10. Subjects with a history (within 2 years of screening) of alcohol abuse that, in the opinion of the Principal Investigator, may impact compliance. Inability to abstain from alcohol consumption during their stay in the hospital/clinic. A positive blood alcohol test at screening is also exclusionary.
11. Any other medical, psychiatric, or social condition that, in the opinion of the investigator, is likely to unfavorably alter the risk-benefit of subject participation, to interfere with protocol compliance, or to confound safety or efficacy assessments.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2028-03-03 (Estimated); Study Completion 2028-03-03 (Estimated)

PRIMARY OUTCOMES:
TEAEs | Through study completion, up to 33 months
  Frequency and severity of TEAEs

SECONDARY OUTCOMES:
SAEs | Through study completion, up to 33 months
  Frequency and severity of serious adverse events (SAEs)
Study Completion | Through study completion, up to 33 months
  Proportion of subjects completing the study
Number of Participants with changes from baseline in safety laboratory values. | Through study completion, up to 33 months
  The number of participants with changes from baseline in the following safety laboratory values: CMP, Hematology (CBC with differential), TSH, Vitamin B12, CRP, Liver Function Test, and Urinalysis will be presented.
Number of Participants with changes from baseline in blood pressure. | Through study completion, up to 33 months
  The number of participants with clinically significant abnormalities in blood pressure from baseline will be presented.
Number of Participants with changes from baseline in heart rate. | Through study completion, up to 33 months
  The number of participants with clinically significant abnormalities in heart rate from baseline will be presented.
Number of Participants with changes from baseline in oxygen saturation. | Through study completion, up to 33 months
  The number of participants with clinically significant abnormalities in oxygen saturation from baseline will be presented.
Number of Participants with changes from baseline in oral temperature. | Through study completion, up to 33 months
  The number of participants with clinically significant abnormalities in oral temperature from baseline will be presented.
Number of Participants with changes from baseline in 12-lead ECG findings. | Through study completion, up to 33 months
  The number of participants with clinically significant abnormalities in 12-lead ECG will be presented. Individual parameters that will be collected include heart rate, PR, QT, QTcF, QRS, and PR intervals.
DTH Response | Through study completion, up to 21 months
  Frequency of a delayed-type hypersensitivity (DTH) response at the ID injection site.
Infusion Reactions | Through study completion, up to 21 months
  Frequency of acute infusion reactions.
Anti-Aβ1-42 antibody titer | Through study completion, up to 33 months
  Evaluation of the anti-Aβ1-42 antibody titer at all collection visits during the study.
Proportion of subjects with anti-Aβ antibodies | Through study completion, up to 33 months
  Proportion of subjects with anti-Aβ antibodies at all collection visits during the study and by visit.
Proportion of subjects with isotype of anti-Aβ antibodies | Through study completion, up to 33 months
  Proportion of subjects with isotype of anti-Aβ antibodies by visit.

CONTACTS AND LOCATIONS:
Locations (1):
- First Excellent Research Group, Doral, Florida, United States

IPD SHARING:
Plan to Share IPD: No